CLINICAL TRIAL: NCT06291545
Title: A Prospective, Multicenter, Randomized Controlled, Non-inferiority Design Clinical Trial, To Evaluate the Efficacy and Safety of the Coronary Artery Notched Balloon Dilation Catheter for the Pre-dilation of Coronary Artery Stenosis Lesions
Brief Title: Effectiveness and Safety of Coronary Scoring Balloon Dilation Catheter in the Pretreatment of Coronary Stenosis Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: JW Medical Systems Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JW-SBC202202
Record Dates: First submitted 2024-02-19; First posted 2024-03-04 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-01

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coronary artery scoring balloon dilation catheter（JW Medical Systems Ltd） (Experimental): Patients with Coronary Artery Disease will be treated with Coronary artery scoring balloon dilation catheter（JW Medical Systems Ltd）
  Interventions: Device: Coronary artery scoring balloon dilation catheter（JW Medical Systems Ltd）
- ScoreFlex NC Coronary Dilatation Catheter (Active Comparator): Patients with Coronary Artery Disease will be treated with ScoreFlex NC Coronary Dilatation Catheter（OrbusNeich Medical [Netherlands] Ltd）
  Interventions: Device: ScoreFlex NC Coronary Dilatation Catheter

INTERVENTIONS:
Device: Coronary artery scoring balloon dilation catheter（JW Medical Systems Ltd） — One hundred subjects who met the inclusion and exclusion criteria were enrolled and assigned to the Coronary artery scoring balloon dilation catheter treatment group.
  Arms: Coronary artery scoring balloon dilation catheter（JW Medical Systems Ltd）
Device: ScoreFlex NC Coronary Dilatation Catheter — One hundred subjects who met the inclusion and exclusion criteria were enrolled and assigned to the ScoreFlex NC Coronary Dilatation Catheter treatment group.
  Arms: ScoreFlex NC Coronary Dilatation Catheter

SUMMARY:
This trial adopts a prospective, multicenter, randomized controlled, and non-inferiority comparison trial design, and plans to recruit 200 eligible subjects who will be randomly assigned to the experimental group or the control group in a 1:1 ratio. All randomly enrolled subjects will be followed up until 30 days after the surgery.

DETAILED DESCRIPTION:
This trial uses a prospective, multicenter, randomized controlled, non-inferiority comparison design. It is expected that the test group will be non-inferior to the control group in the main effectiveness evaluation index (device success rate). This trial plans to enroll 200 subjects who meet the requirements, and they will be randomly assigned to the test group or the control group in a 1:1 ratio. All randomly enrolled subjects will be followed up for 30 days after percutaneous coronary intervention (PCI) treatment to compare the test group and the control group in the main effectiveness evaluation index (device success rate), secondary effectiveness evaluation indices (immediate lumen gain [QCA analysis], surgical success rate, in-hospital major adverse cardiac event [MACE] incidence rate, target lesion failure [TLF] incidence rate within 30 days after surgery, patient-related composite endpoints [PoCE] incidence rate during and within 30 days after surgery, device operation and performance evaluation), and safety evaluation indices (device-related complication incidence rate, adverse event/serious adverse event incidence rate, device defect incidence rate), in order to evaluate the effectiveness and safety of the coronary scoring balloon dilation catheter of the test medical device.

ELIGIBILITY:
Inclusion Criteria:

* 1. Voluntary participation in this trial and signed the informed consent form;
* 2. Age: ≥18 and ≤80 years old, regardless of gender;
* 3. The existence of coronary artery stenosis lesions accompanied by evidence of ischemia in the heart (such as symptomatic coronary heart disease, stable/unstable angina pectoris or asymptomatic myocardial ischemia), suitable for percutaneous interventional therapy.

Exclusion Criteria:

* 1. Acute myocardial infarction (AMI) within 7 days before surgery;
* 2. Serum creatinine level >2.0 mg/dL (177 umol/L) within 7 days before surgery;
* 3. Active peptic ulcer or active gastrointestinal bleeding within 1 month before surgery;
* 4. Stroke or transient ischemic attack (TIA) within 3 months before surgery;
* 5. Known left ventricular ejection fraction (LVEF) <30% (if LVEF is unknown, it can be measured during this surgery);
* 6. Known allergies to aspirin or heparin or the existence of contraindications that prevent the subjects from receiving sufficient preoperative medications;
* 7. Known subjects allergic to ingredients in the test product or contrast agent;
* 8. Known subjects who are pregnant or breastfeeding;
* 9. Planned to use coronary atherectomy, laser ablation, other scoring / spiked / cutting balloons (non-study devices) or shock wave balloons to treat the target lesion at the same time;
* 10. Subjects participating in other drug or device clinical studies;
* 11. Other situations that are not suitable for participation in this study as assessed by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-03-20 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Rate of successful device usage | 1hour
  The investigational device was successfully delivered to the intended target lesion, dilated, deflated, and retrieved smoothly; After balloon angioplasty with the investigational device, the residual stenosis of the target lesion diameter was <50%.

SECONDARY OUTCOMES:
Rate of success of the surgery | 3 days
  The success of the surgery is defined as on the basis of successful use of the instrument, the residual stenosis of the target lesion diameter after PCI is ≤ 30% and TIMI blood flow is grade 3, and no MACE occurs in the hospital.
Incidence of in-hospital MACE | 30 days
  MACE includes cardiac death, target vessel myocardial infarction, and target lesion re-vascularization
Incidence of PoCE within 30 days after surgery | 30 days
  PoCE includes all-cause mortality, all MIs, and any re-vascularization
The lumen is obtained immediately | 1hour
  The lumen is obtained immediately (QCA analysis)

CONTACTS AND LOCATIONS:
Overall Officials: Ling Tao, Ph.D, Principal Investigator — The First Affiliated Hospital of Air Force Medical University

IPD SHARING:
Plan to Share IPD: No